CLINICAL TRIAL: NCT03228238
Title: Effects of Long-term Vitamin C+E and Statin Therapy on Vasospasm Improvement and Regression of Atheroma in Patients With Variant Angina
Brief Title: ANti-Oxidant in Variant Angina (ANOVA) Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Director of Cardiac Catheterization Laboratory & Coronary Intervention, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANOVA
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Variant Angina
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — Ascorbic Acid; Vitamin E; Tocopherols; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Calcium Channel Blockers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dual subgroup (Experimental): Standard medication for variant angina plus Vitamin C+E plus Statin Vitamin C and Vitamin E : Ascorbic acid Tablet 1g / Tocopherol Capsule 400IU Statin : Atorvastatin calcium 10mg
  Interventions: Drug: Vitamin C and Vitamin E; Drug: Statin; Drug: Standard medication for variant angina
- Statin subgroup (Experimental): Standard medication for variant angina plus Statin Statin : Atorvastatin calcium 10mg
  Interventions: Drug: Statin; Drug: Standard medication for variant angina
- Vitamin subgroup (Experimental): Standard medication for variant angina plus Vitamin C+E Vitamin C and Vitamin E : Ascorbic acid Tablet 1g / Tocopherol Capsule 400IU
  Interventions: Drug: Vitamin C and Vitamin E; Drug: Standard medication for variant angina
- Control group (Active Comparator): Control subgroup : Standard medication for Variant angina only
  Interventions: Drug: Standard medication for variant angina

INTERVENTIONS:
Drug: Vitamin C and Vitamin E — Ascorbic acid Tablet 1g and Tocopherol Capsule 400IU
  Other Names: Ascorbic acid and Tocopherol
  Arms: Dual subgroup; Vitamin subgroup
Drug: Statin — Atorvastatin calcium 10mg
  Other Names: Atorvastatin
  Arms: Dual subgroup; Statin subgroup
Drug: Standard medication for variant angina — Calcium Channel blocker or NG
  Other Names: Calcium Channel blocker or NG

SUMMARY:
Purpose Objectives

1. To evaluate the anti-oxidant effect of long-term Vitamin C+E therapy on coronary vasospasm improvement.
2. To evaluate the anti-oxidant effect of long-term statin therapy on coronary vasospasm improvement.
3. To evaluate the effect of long-term Vitamin C+E and statin therapy on regression of atheroma in target coronary vessels via intravascular ultrasound.
4. To find out the role of vascular endothelium in variant angina via evaluating long-term Vitamin C+E and statin therapy on improvement in vascular endothelial function by assessing brachial arterial expansion capability.
5. To find out the role of vascular endothelium in variant angina via evaluating long-term Vitamin C+E and statin therapy on improvement in arterial stiffness by assessing pulse wave velocity(PWV)

DETAILED DESCRIPTION:
Study Design: Prospective, open label, Four-arm, randomized single-center trial to test the effect long-term Vitamin C+E and Statin therapy on vasospasm improvement and regression of atheroma in patients with variant angina.

After provocation test, patients will be classified into three groups.(See below)

1. Negative group : Patients who have symptoms that are consistent with vasospastic angina but only show luminal narrowing less than 50% on coronary angiography during provocation test.
2. Mild Spastic group : Patients who have symptoms that are consistent with vasospastic angina and show luminal narrowing over 50% to less than 90% on coronary angiography during provocation test.
3. Severe Spastic group : Patients who have symptoms that are consistent with vasospastic angina and show luminal narrowing over 90% on coronary angiography during provocation test.

In each group (except for patient in Negative group), patients will be randomized in a two by two factorial manner according to the study drug therapy (Vitamin C+E vs. no Vitamin C+E) (Statin vs. no Statin) As a result, patients in each group(except for patient in Negative group) will be randomized to 4 treatment subgroups, which are

1. Control subgroup : Standard medication for Variant angina only
2. Vitamin subgroup : Standard medication + Vitamin C+E
3. Statin subgroup : Standard medication + Statin
4. Dual subgroup : Standard medication + Vitamin C+E + Statin

Patients in Negative group will be prescribed only for standard medication for variant angina.

Patient Enrollment: Recruiting 300 patients(100 patients for each group, as 25 patients for each subgroups) from September 2014 through February 2021 at single center in Korea(Seoul National University Hospital)

Patient Follow-Up: Clinical follow-up will occur at 1, and 6 months, and at 2, 4, and 6 years. Investigator or designee may conduct follow-up as telephone contacts or office visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 30 years of age.
2. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the Vitamin C+E or Statin or Dual, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
3. Subject must have symptoms that are consistent with vasospastic angina with planned Coronary angiography and Provocation test.

Exclusion Criteria:

1. Patient who has organic coronary stenosis in main coronary branch at least 50% luminal narrowing after intracoronary nitroglycerin injection
2. Patient who has continuously taken Vitamin C or Vitamin E or Statin within 3months before Admission
3. Creatinine level ≥ 2.0mg/dL or dependence on dialysis.
4. Severe hepatic dysfunction (AST and ALT: 3 times upper normal reference values).
5. Active Myopathy or elevated Creatine kinase enzyme level (3 times upper normal reference values).
6. History of Severe hepatic dysfunction or Rhabdomyolysis due to statin side effect
7. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
8. History of Urolithiasis
9. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Vasospasm at 6months | at 6 months
  Severity of vasospasm in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to control subgroup.
Vasospasm at 2 years | at 2 years
  Severity of vasospasm in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to control subgroup.
Vasospasm at 4 years | at 4 years
  Severity of vasospasm in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to control subgroup.
Vasospasm at 6 years | at 6 years
  Severity of vasospasm in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to control subgroup.

SECONDARY OUTCOMES:
Changes from baseline in Vasospasm | at 6 months, and at 2, 4, and 6 years follow up period
  Changes of Vasospasm in Control subgroup, Vitamin subgroup, Statin subgroup, and Dual subgroup compared to baseline vasospasm assessed by provocation test.
Composed improvement of Vascular endothelial function(Brachial arterial expansion capability) | at 6 months, and at 2, 4, and 6 years follow up period
  in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to control subgroup
Improvement of Vascular endothelial function(Brachial arterial expansion capability) | at 6 months, and at 2, 4, and 6 years follow up period
  in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to baseline endothelial function test results
Comparative analysis of improvement of Vascular endothelial function(Brachial arterial expansion capability) | at 6 months, and at 2, 4, and 6 years follow up period
  in Vitamin subgroup, Statin subgroup, and Dual subgroup
Composed improvement of Arterial stiffness(Pulse wave velocity(PWV)) | at 6 months, and at 2, 4, and 6 years follow up period
  in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to control subgroup
Improvement of Arterial stiffness(Pulse wave velocity(PWV)) | at 6 months, and at 2, 4, and 6 years follow up period
  in Vitamin subgroup, Statin subgroup, and Dual subgroup compared to baseline endothelial function test results
Comparative analysis of improvement of Arterial stiffness(Pulse wave velocity(PWV)) | at 6 months, and at 2, 4, and 6 years follow up period
  in Vitamin subgroup, Statin subgroup, and Dual subgroup

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea